CLINICAL TRIAL: NCT01148511
Title: Comparison of Safety, Effectiveness, and Quality-of-life Outcomes Between Labeled Versus "Treat and Extend" Regimen in Turkish Patients With Choroidal Neovascularisation Due to AMD
Brief Title: Comparison of Safety, Effectiveness and Quality of Life Outcomes Between Labeled Versus "Treat and Extend" Regimen in Turkish Patients With Choroidal Neovascularisation Due to Age-related Macular Degeneration (AMD)
Acronym: SALUTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002ATR01
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Age-related Macular Degeneration
Keywords: Macula degeneration; Ranibizumab; Choroidal neovascularisation; Treat and extend; Treat and observe
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Ranibizumab

ARMS (2):
- Treat and Extend (Experimental): Patients received ranibizumab 0.5 mg intravitreally (ivt) once a month for 3 months. If the disease was inactive 4 weeks later, the next visit was postponed 2 weeks to 6 weeks later. If the disease was inactive during subsequent visits, the next visit was postponed an additional 2 weeks to 8 weeks later, the maximum interval between visits. If the disease became active at any visit, the patient received ranibizumab 0.5 mg ivt and the follow-up schedule started over.
  Interventions: Drug: Ranibizumab 0.5 mg
- Treat and Observe (Active Comparator): Patients received ranibizumab 0.5 mg intravitreally (ivt) once a month for 3 months. All subsequent visits occurred monthly. If the disease was active, the patient received ranibizumab 0.5 mg ivt. If the disease was inactive, no treatment was administered and the patient was instructed to return 1 month later.
  Interventions: Drug: Ranibizumab 0.5 mg

INTERVENTIONS:
Drug: Ranibizumab 0.5 mg — Ranibizumab was supplied as a sterile solution in sealed glass vials.
  Other Names: Lucentis

SUMMARY:
The purpose of the study was to compare 2 treatment regimens for patients suffering from choroidal neovascularisation secondary to age-related macular degeneration (AMD). The first treatment regimen was the approved AMD treatment of 1 injection each month for 3 months and than re-treatment of patients who have a visual loss of more than 5 letters with monthly control (Treat and Observe). The second treatment regimen was 1 injection each month for 3 months and than extending the control period if the macula is dry during the monthly control (Treat and Extend). If the "Treat and Extend" regimen is found effective and safe, the number of ranibizumab injections, the number of patient visits, the risk of adverse events due to the intravitreal injections, and policlinic occupation number could all be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over the age of 50.
* Patients with primary, secondary, or recurrent subfoveal choroidal neovascularization (CNV) to AMD with classic, minimal classic, or occult lesions.
* Patients with CNV area ≥ %50 of the total lesion.
* Total lesion area ≤ 12 disc areas for minimal classic/occult lesions and ≤ 9 disc areas for the classic lesions.
* Best-corrected visual acuity (BCVA) score between 73 and 34 letters in the study eye.

Exclusion Criteria:

* BCVA < 34 letters.
* Patients using anti-angiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, corticosteroids, or protein kinase C inhibitors, etc) or inclusion in another trial (for any eye).
* Verteporphin, external radiational therapy, subfoveal focal laser photocoagulation, vitrectomy, or transpupillary thermotherapy application to the eye before the study.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Turkey (Türkiye) (8):
  - Novartis Investigative Site, Adana
  - Novartis Investigational Site, Ankara
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Bursa
  - Novartis Investigative Site, Eskişehir
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Konya

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All 99 patients were exposed to study drug. 93 of the 99 patients were randomized into the Treat and Extend and the Treat and Observe treatment groups.
Period: Exposed to Study Drug
Arm/Group | All Patients | Treat and Extend | Treat and Observe
Started | 99 | 0 (Patients were not randomized to this group until the Randomized Period.) | 0 (Patients were not randomized to this group until the Randomized Period.)
Completed | 93 | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Period: Randomized
Arm/Group | All Patients | Treat and Extend | Treat and Observe
Started | 0 (All patients were randomized into the Treat and Extend and the Treat and Observe treatment groups.) | 48 | 45
Completed | 0 | 38 | 39
Not Completed | 0 | 10 | 6
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Consent withdrawal | 0 | 5 | 3
Not completed — Other | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: All patients who received study drug (n=99). Not all patients who received study drug were randomized into the 2 treatment groups (n=93) due to discontinuation from the study in the first Period of the study. Baseline Characteristics are only reported for the randomized (n=93) patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treat and Extend | Treat and Observe | Total
Number analyzed (Participants) | 48 | 45 | 93
Age Continuous [Mean (Standard Deviation); unit: years] | 70.8 (8.8) | 71.1 (8.4) | 70.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Best-Corrected Visual Acuity (logMAR) From Baseline to Month 12
Description: Best corrected visual acuity (BCVA) was assessed in the study eye. BCVA measurements were made using the logarithm of the minimum angle of resolution (logMAR) visual acuity testing charts. Each letter on the chart has a score value of 0.02 log units. Since there are 5 letters per line, the total score for a line on the logMAR chart represents a change of 0.1 log units. The formula for calculating the logMAR BCVA score is: 0.1 + logMAR value of the best line read - 0.02 x number of letters read. A lower BCVA score indicates better vision. A negative change score indicates improvement.
Time Frame: Baseline to Month 12
Population: Per protocol population: All patients who were evaluated at Baseline and at 12±2 months. Patients who discontinued from the study were not included in the per protocol population.
Measure: Median (Full Range); unit: logMAR
Arm/Group | Treat and Extend | Treat and Observe
Number analyzed (Participants) | 38 | 39
logMAR | -0.18 [-0.88 to 0.76] | -0.12 [-0.88 to 1.56]

2. Primary Outcome: Change in Letter Count From Baseline to Month 12
Description: Letter count was assessed in the study eye. Measurements were made using the logarithm of the minimum angle of resolution (logMAR) visual acuity testing charts. A higher letter count score indicates better vision. A negative change score indicates improvement.
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Letters
Arm/Group | Treat and Extend | Treat and Observe
Number analyzed (Participants) | 38 | 39
Letters | -9 [-44 to 38] | -6 [-44 to 78]

3. Secondary Outcome: Letter Count From Baseline to Month 12
Description: Letter count was assessed in the study eye. Measurements were made using the logarithm of the minimum angle of resolution (logMAR) visual acuity testing charts. Results are reported in various categories of change in letter count.
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Treat and Extend | Treat and Observe
Number analyzed (Participants) | 38 | 39
Percentage of patients
  < 35 letters | 7.9 | 7.7
  ≥ 35 letters | 92.1 | 92.3
  loss > 15 letters | 10.5 | 10.3
  loss ≤ 15 letters or gained letter | 89.5 | 89.7
  loss ≥ 30 letters | 2.6 | 5.1
  loss < 30 letters or gained letter | 97.4 | 94.9
  gain ≥ 0 letter | 76.3 | 61.5
  Loss | 23.7 | 38.5
  gain ≥ 15 letter | 34.2 | 23.1
  gain < 15 letters or loss | 65.8 | 76.9

4. Secondary Outcome: Number of Visits
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Visits
Arm/Group | Treat and Extend | Treat and Observe
Number analyzed (Participants) | 38 | 39
Visits | 12.0 [10.0 to 15.0] | 15.0 [12.0 to 15.0]

5. Secondary Outcome: Follow-up Duration
Description: Follow-up duration was defined as the number of days from Baseline to study discontinuation.
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Mean (Full Range); unit: Days
Arm/Group | Treat and Extend | Treat and Observe
Number analyzed (Participants) | 38 | 39
Days | 364.5 [310.0 to 396.0] | 366.0 [320.0 to 386.0]

6. Secondary Outcome: Change in Central Retinal Thickness From Baseline to Month 12
Description: Retinal thickness was measured using Optical Coherence Tomography (OCT).
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Median (Full Range); unit: µm
Arm/Group | Treat and Extend | Treat and Observe
Number analyzed (Participants) | 38 | 39
µm | 88.5 [-190.0 to 584.0] | 61.0 [-470.0 to 500.0]

7. Secondary Outcome: Quality of Life
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) was used to measure a patient's subjective assessment of vision-related quality of life at Visits 2, 6, 9, 12, and 15. The 12 subscales in the VFQ-25 are general health, general vision, ocular pain, near activities, distance activities, social function, mental health, role difficulties, dependency, driving, color vision, and peripheral vision. The scores on the subscales were added together for a total score, which ranged from 0 to 100. A higher score indicated poorer function.
Time Frame: Visits 2, 6, 9, 12, and 15 (up to 12 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Treat and Extend | Treat and Observe
Number analyzed (Participants) | 27 | 30
Units on a scale
  Visit 2 | 70.0 [57.0 to 87.0] | 73.0 [62.0 to 89.0]
  Visit 6 | 71.0 [65.0 to 83.0] | 69.5 [60.0 to 79.0]
  Visit 9 | 69.0 [63.0 to 80.0] | 72.5 [62.0 to 92.0]
  Visit 12 | 72.0 [64.0 to 84.0] | 71.0 [60.0 to 91.0]
  Visit 15 | 69.0 [64.0 to 80.0] | 70.5 [57.0 to 85.0]

ADVERSE EVENTS:
Description: Safety population: All patients who received study drug.
Groups:
- Before Randomization: These 6 patients were exposed to study drug but discontinued from the study prior to randomization.
Arm/Group | Treat and Extend | Treat and Observe | Before Randomization
Serious Adverse Events (participants affected / at risk) | 5/48 | 3/45 | 2/6
Other Adverse Events (participants affected / at risk) | 10/48 | 8/45 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treat and Extend (N=48) | Treat and Observe (N=45) | Before Randomization (N=6)
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Lower and upper limb fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Aphasia Syncope (Psychiatric disorders) | 0 | 1 | 0
Azotemia (Renal and urinary disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vascular graft (Surgical and medical procedures) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treat and Extend (N=48) | Treat and Observe (N=45) | Before Randomization (N=6)
Adenoviral conjunctivitis (Eye disorders) | 2 | 3 | 0
Influenza (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.